CLINICAL TRIAL: NCT04217785
Title: Umbilical Cord Serum Versus Conventional Eyedrops In Treatment of Moderate To Severe Dry Eye Disease: A Randomized Clinical Trial
Brief Title: Umbilical Cord Serum Versus Conventional Eyedrops
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Wan Haslina Wan Abdul Halim, Consultant Ophthalmologist-Cornea And Anterior Segment, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FF-2019-209; GGPM-2018-052 (Other Grant/Funding Number: National University of Malaysia)
Record Dates: First submitted 2019-12-23; First posted 2020-01-03 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Dry Eye Syndromes
Keywords: Umbilical Cord Serum Eyedrops; Moderate To Severe Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-AT eye drops (Active Comparator): Optive Fusion UD eye drops + Genteal lubricant gel
  Interventions: Drug: Optive, Ophthalmic Solution; Drug: Genteal lubricant gel
- B-UCS eye drops (Active Comparator): UCS eye drops + GentTeal lubricant gel
  Interventions: Biological: Umbilical Cord Serum eye drops; Drug: Genteal lubricant gel

INTERVENTIONS:
Drug: Optive, Ophthalmic Solution — 6 drops per day, for 8 weeks
  Other Names: Optive Fusion UD
  Arms: A-AT eye drops
Biological: Umbilical Cord Serum eye drops — UCS eye drops (6 drops per day, for 8 weeks)
  Arms: B-UCS eye drops
Drug: Genteal lubricant gel — Genteal lubricant gel (2 drops per day, for 8 weeks)

SUMMARY:
Dry eye disease (DED) is a chronic ocular surface disease and the prevalence of DED has been reported as high as 50%. Recently, The international Dry Eyes Workshop II (DEWS II) defines dry eye as a "multifactorial disease of the ocular surface characterized by a loss of homeostasis of the tear film, and accompanied by ocular symptoms, in which tear film instability and hyperosmolarity, ocular surface inflammation and damage, and neurosensory abnormalities play etiological roles". A study done by Yoon et al. on 31 patients with severe DED concluded that UCS eye drops are effective and safe in treating severe DED. Studies found that EGF, TGF-β, VEGF and vitamin A levels were significantly higher in UCS than peripheral blood serum(PBS) whereas IGF content was significantly higher in PBS than in CBS. Yoon et al. then conducted another study whereby he compared UCS to AS in treating both Sjögren syndrome and non- Sjögren syndrome patients with severe dry eyes. They concluded that UCS eye drops were more effective in decreasing symptoms and keratoepitheliopathy in severe dry eye syndrome and increasing goblet cell density in Sjögren syndrome compared with AS drops. Despite proven more effective in treating DED, serum eye drops are not yet widely manufactured due to a few reasons. This study is chosen because

1. Not many previous clinical trials done related to UCS eye drops.
2. There were only two clinical trials done before to compare the use of UCS eye drops versus conventional AT eye drops on Hansen's disease and acute ocular chemical burn injury population.
3. To apply the newer technology of Keratograph® 5M in DED assessment.
4. To initiate a proper standard operating procedure for production as well as delivery of serum eye drops which allowing out-patient treatment with serum eye drops possible.

DETAILED DESCRIPTION:
This is a prospective, single- blinded randomized clinical trial conducted in University Kebangsaan Malaysia Medical Centre (UKMMC). Umbilical cord serum will be provided by Pusat Darah Negara (National Blood Centre), Malaysia. All patients from Ophthalmology Clinic in UKM Medical Centre from December 2019 till December 2021 will be involved in this study. Patients who fulfill the inclusion criteria will be included in this study. Informed consent will be taken and dry eye assessment that includes visual acuity, OSDI score, Schirmer test, NITBUT, corneal fluorescein staining, TMH and conjunctival injection. The patients will be randomised into 2 groups; AT eye drops and UCS eye drops.

Human umbilical cord blood samples will be collected from Maternity Hospital, Hospital Kuala Lumpur with assistance of the nurses from Cord Blood Collection Unit. All maternal blood samples were collected after the written informed consent from respective parents and subjected for virology screening.

National Blood Bank has a procedure for virology screening and all collected maternal umbilical cord bloods will be screened for Hep B Surface Antigen, Anti-HCV Ag/Ab, HIV Ag/Ab, Syphillis and Cytomegalovirus (CMV) IgM in Transfusion Microbiology Laborator (Accredited by ISO 15189 and CSL). Method that has been used in the screening as below:

* Hep B Surface Antigen, Anti-HCV, HIV Ag/Ab: Chemiluminescent Microparticle Immunoassay (CMIA).
* Syphilis : Carbon Antigen (Manual)
* CMV IgM : Electrochemiluminescence Immunoassay (ECLIA)

Whereas, the CB samples are screened for bacteriology screening pre and post processing to ensure sterility of the product. The serum will be discarded if any of the laboratory results are positive or reactive.

The collected cord blood (CB) will then be placed in an incubator at the collection centre until the cord blood samples are sent to National Blood Bank in an ice box with temperature logger. Once the ice box reached National Blood Bank, MLT will check the temperature logger and make sure all the temperature data within range (10-26oC) before starting the UCS serum eye drops production.

CB will be processed in Cord Blood Processing Unit within 24 hours of collection to ensure retrieval of high quality of bioactive molecules. Laboratory temperature room, humidity and oxygen will be monitored twice a day. Upon arrival at the processing laboratory, the CB will then be left at room temperature for about 2 hours to allow the CB to clot completely. After 15 minutes of centrifugation at 3,000 × g, under sterile conditions, the serum fraction will be carefully separated from the cellular fraction. Separated serum is then transferred to a tygon tube by using a sterile docking device and diluted to a 20% dilution with balanced salt solution (BSS) without any antibiotics, and finally sealed into 1-inch segment consisting of approximately 1 ml serum eye drops. The segmented UCS will then be frozen at -20oC for 3 to 6 months or at -80°C for long term storage.

For safety and quality interest, frozen segments will be transported to UKMMC blood bank using a transportation box filled with dry ice to ensure UCS are at frozen state and to maintain the quality of the product until they reach destination. From UKMMC blood bank, participants will need to bring the frozen UCS eye drops home by transporting them in a cooler box with ice packs. At home, the frozen UCS eye drops will need to be kept in domestic freezer. The frozen UCS eye drops must be thawed at room temperature prior to usage and thereafter stored in the refrigerator at 2-8°C for a maximum of 24 hours. A short instruction sheet will be provided to participants on UCS usage. There will be no porcine/bovine materials involved in the whole process.

Statistical analysis will be performed using Statistical Package for Social Science, version 20.0 (SPSS, Inc., Chicago, III., USA) for Windows. Mean value comparisons between study groups can be performed with the Student's T-test using 2 sided-analysis. Mean value comparisons for follow up can be analysed with ANOVA. Categorical characteristics can be analyzed using a Chi-square. Differences are considered statistically significant at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Dry Eye Disease based on OSDI score or DED severity grading scheme
* Patients willing to participate in this study and able to provide consent
* Patients with domestic freezer at home

Exclusion Criteria:

* Infective cases
* Cases with limbal stem cells deficiency
* Patients with lid abnormalities
* Allergic to study eye drops component

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of change in corneal surface in patients treated with Umbilical Cord Serum eyedrops and conventional AT eyedrops | At 4th week of treatment
  Change of non-invasive tear break-up time (s) and Tear Break-up Time (s) of corneal surface from Baseline by using Oculus Keratograph-5 Machine at 4th week of eyedrop instillation.
Comparison of change in corneal surface in patients treated with Umbilical Cord Serum eyedrops and conventional AT eyedrops | At 8th week of treatment
  Change of non-invasive tear break-up time (s) and Tear Break-up Time (s) of corneal surface from Baseline by using Oculus Keratograph-5 Machine at 8th week of eyedrop instillation.
Comparison of meniscometry (mm) in patients treated with Umbilical Cord Serum eyedrops and conventional AT eyedrops | At 4th week of treatment
  Change in tear meniscus height (mm) of corneal surface from Baseline by using Oculus Keratograph-5 Machine at 4th week of eyedrop instillation.
Comparison of meniscometry (mm) in patients treated with Umbilical Cord Serum eyedrops and conventional AT eyedrops | At 8th week of treatment
  Change in tear meniscus height (mm) of corneal surface from Baseline by using Oculus Keratograph-5 Machine at 8th week of eyedrop instillation.
Comparison of change in corneal surface signs in patients treated with Umbilical Cord Serum eyedrops and conventional AT eyedrops | At 4th week of treatment
  Change of Corneal surface signs (ie punctate epithelial erosions) from Baseline based on Oxford Scale Eye Grading through slit-lamp examination at 4th week of eyedrop instillation. The grade ranges from 0-5, in which higher scores indicate worse outcome.
Comparison of change in corneal surface signs in patients treated with Umbilical Cord Serum eyedrops and conventional AT eyedrops | At 8th week of treatment
  Change of Corneal surface signs (ie punctate epithelial erosions) from Baseline based on Oxford Scale Eye Grading through slit-lamp examination at 8th week of eyedrop instillation. The grade ranges from 0-5, in which higher scores indicate worse outcome.
Comparison of ocular surface redness in patients treated with Umbilical Cord Serum eyedrops and conventional AT eyedrops | At 4th week of treatment
  Change of ocular surface redness from Baseline based on Redness Scoring using Oculus Keratograph-5 Machine at 4th week of eyedrop instillation.
Comparison of ocular surface redness in patients treated with Umbilical Cord Serum eyedrops and conventional AT eyedrops | At 8th week of treatment
  Change of ocular surface redness from Baseline based on Redness Scoring using Oculus Keratograph-5 Machine at 8th week of eyedrop instillation.
Comparison of change in basal tear production in patients treated with Umbilical Cord Serum eyedrops and conventional AT eyedrops | At 4th week of treatment
  Change of basal tear production (mm) from Baseline through Schirmer's test at 4th week of eyedrop instillation.
Comparison of change in basal tear production in patients treated with Umbilical Cord Serum eyedrops and conventional AT eyedrops | At 8th week of treatment
  Change of basal tear production (mm) from Baseline through Schirmer's test at 8th week of eyedrop instillation.
Comparison of dry eye symptom improvements in patients treated with Umbilical Cord Serum eyedrops and conventional AT eyedrops | At 4th week of treatment
  Change of dry eye symptoms from baseline based on Ocular Surface Disease Index (OSDI) score at 4th week of eyedrop instillation.
Comparison of dry eye symptom improvements in patients treated with Umbilical Cord Serum eyedrops and conventional AT eyedrops | At 8th week of treatment
  Change of dry eye symptoms from baseline based on Ocular Surface Disease Index (OSDI) score at 8th week of eyedrop instillation.

CONTACTS AND LOCATIONS:
Overall Officials: Wan Haslina Wan Abdul Halim, M.D(UKM), Study Chair — National University of Malaysia
Locations (3):
- Malaysia (3):
  - UKM Medical Centre, Cheras, Kuala Lumpur
  - National Blood Centre, Malaysia, Kuala Lumpur, Kuala Lumpur
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur

REFERENCES:
- [Background] Lemp MA. Report of the National Eye Institute/Industry workshop on Clinical Trials in Dry Eyes. CLAO J. 1995 Oct;21(4):221-32. No abstract available. PMID 8565190
- [Background] Aggarwal S, Kheirkhah A, Cavalcanti BM, Cruzat A, Colon C, Brown E, Borsook D, Pruss H, Hamrah P. Autologous Serum Tears for Treatment of Photoallodynia in Patients with Corneal Neuropathy: Efficacy and Evaluation with In Vivo Confocal Microscopy. Ocul Surf. 2015 Jul;13(3):250-62. doi: 10.1016/j.jtos.2015.01.005. Epub 2015 Feb 20. PMID 26045233
- [Background] The definition and classification of dry eye disease: report of the Definition and Classification Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):75-92. doi: 10.1016/s1542-0124(12)70081-2. PMID 17508116
- [Background] Bradley JC, Simoni J, Bradley RH, McCartney DL, Brown SM. Time- and temperature-dependent stability of growth factor peptides in human autologous serum eye drops. Cornea. 2009 Feb;28(2):200-5. doi: 10.1097/ICO.0b013e318186321e. PMID 19158565
- [Background] Bron AJ, de Paiva CS, Chauhan SK, Bonini S, Gabison EE, Jain S, Knop E, Markoulli M, Ogawa Y, Perez V, Uchino Y, Yokoi N, Zoukhri D, Sullivan DA. TFOS DEWS II pathophysiology report. Ocul Surf. 2017 Jul;15(3):438-510. doi: 10.1016/j.jtos.2017.05.011. Epub 2017 Jul 20. PMID 28736340
- [Background] Celebi AR, Ulusoy C, Mirza GE. The efficacy of autologous serum eye drops for severe dry eye syndrome: a randomized double-blind crossover study. Graefes Arch Clin Exp Ophthalmol. 2014 Apr;252(4):619-26. doi: 10.1007/s00417-014-2599-1. Epub 2014 Feb 25. PMID 24566903
- [Background] Chiang CC, Lin JM, Chen WL, Tsai YY. Allogeneic serum eye drops for the treatment of severe dry eye in patients with chronic graft-versus-host disease. Cornea. 2007 Aug;26(7):861-3. doi: 10.1097/ICO.0b013e3180645cd7. PMID 17667623
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Dietrich T, Weisbach V, Seitz B, Jacobi C, Kruse FE, Eckstein R, Cursiefen C. [Manufacture of autologous serum eye drops for out-patient therapy : cooperation between ophthalmic clinic and transfusion medicine department]. Ophthalmologe. 2008 Nov;105(11):1036-8, 1040-2. doi: 10.1007/s00347-008-1692-4. German. PMID 18506408
- [Background] Esquenazi S, He J, Bazan HE, Bazan NG. Use of autologous serum in corneal epithelial defects post-lamellar surgery. Cornea. 2005 Nov;24(8):992-7. doi: 10.1097/01.ico.0000160967.65953.ea. PMID 16227849
- [Background] Farrand KF, Fridman M, Stillman IO, Schaumberg DA. Prevalence of Diagnosed Dry Eye Disease in the United States Among Adults Aged 18 Years and Older. Am J Ophthalmol. 2017 Oct;182:90-98. doi: 10.1016/j.ajo.2017.06.033. Epub 2017 Jul 10. PMID 28705660
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Foulks, G., Lemp, M., Jester, J., Sutphin, J., Murube, J. & Novack, G. 2007. Report of the International Dry Eye Workshop (Dews). Ocul Surf 5(2): 65-204.
- [Background] Guo B, Lu P, Chen X, Zhang W, Chen R. Prevalence of dry eye disease in Mongolians at high altitude in China: the Henan eye study. Ophthalmic Epidemiol. 2010 Aug;17(4):234-41. doi: 10.3109/09286586.2010.498659. PMID 20642346
- [Background] Hussain M, Shtein RM, Sugar A, Soong HK, Woodward MA, DeLoss K, Mian SI. Long-term use of autologous serum 50% eye drops for the treatment of dry eye disease. Cornea. 2014 Dec;33(12):1245-51. doi: 10.1097/ICO.0000000000000271. PMID 25299423
- [Background] Jirsova K, Brejchova K, Krabcova I, Filipec M, Al Fakih A, Palos M, Vesela V. The application of autologous serum eye drops in severe dry eye patients; subjective and objective parameters before and after treatment. Curr Eye Res. 2014 Jan;39(1):21-30. doi: 10.3109/02713683.2013.824987. Epub 2013 Sep 27. PMID 24074049
- [Background] Jones L, Downie LE, Korb D, Benitez-Del-Castillo JM, Dana R, Deng SX, Dong PN, Geerling G, Hida RY, Liu Y, Seo KY, Tauber J, Wakamatsu TH, Xu J, Wolffsohn JS, Craig JP. TFOS DEWS II Management and Therapy Report. Ocul Surf. 2017 Jul;15(3):575-628. doi: 10.1016/j.jtos.2017.05.006. Epub 2017 Jul 20. PMID 28736343
- [Background] Kojima T, Ishida R, Dogru M, Goto E, Matsumoto Y, Kaido M, Tsubota K. The effect of autologous serum eyedrops in the treatment of severe dry eye disease: a prospective randomized case-control study. Am J Ophthalmol. 2005 Feb;139(2):242-6. doi: 10.1016/j.ajo.2004.08.040. PMID 15733983
- [Background] Lemp MA, Crews LA, Bron AJ, Foulks GN, Sullivan BD. Distribution of aqueous-deficient and evaporative dry eye in a clinic-based patient cohort: a retrospective study. Cornea. 2012 May;31(5):472-8. doi: 10.1097/ICO.0b013e318225415a. PMID 22378109
- [Background] Lopez-Garcia JS, Garcia-Lozano I, Rivas L, Gimenez C, Acera A, Suarez-Cortes T. Effects of Autologous Serum Eye Drops on Conjunctival Expression of MUC5AC in Patients With Ocular Surface Disorders. Cornea. 2016 Mar;35(3):336-41. doi: 10.1097/ICO.0000000000000726. PMID 26785302
- [Background] Moh, M. O. H. M. 2009. Keputusan Muzakarah Jawatankuasa Fatwa Majlis Kebangsaan Bagi Hal Ehwal Agama Islam Malaysia Berkaitan Pengklonan Dan Art. 2nd Edition Malaysian Guidelines for Stem Cell Research and Therapy
- [Background] Noble BA, Loh RS, MacLennan S, Pesudovs K, Reynolds A, Bridges LR, Burr J, Stewart O, Quereshi S. Comparison of autologous serum eye drops with conventional therapy in a randomised controlled crossover trial for ocular surface disease. Br J Ophthalmol. 2004 May;88(5):647-52. doi: 10.1136/bjo.2003.026211. PMID 15090417
- [Background] Noda-Tsuruya T, Asano-Kato N, Toda I, Tsubota K. Autologous serum eye drops for dry eye after LASIK. J Refract Surg. 2006 Jan-Feb;22(1):61-6. doi: 10.3928/1081-597X-20060101-13. PMID 16447938
- [Background] Rahman, A. a. A., Badarudin, N. E., Azemin, M. Z. C. & Ariffin, A. E. 2017. Development of a Bahasa Melayu Version of Ocular Surface Disease Index (Osdi). INTERNATIONAL JOURNAL OF ALLIED HEALTH SCIENCES 1(1):
- [Background] Ralph RA, Doane MG, Dohlman CH. Clinical experience with a mobile ocular perfusion pump. Arch Ophthalmol. 1975 Oct;93(10):1039-43. doi: 10.1001/archopht.1975.01010020815015. PMID 1180750
- [Background] Uchino M, Schaumberg DA. Dry Eye Disease: Impact on Quality of Life and Vision. Curr Ophthalmol Rep. 2013 Jun;1(2):51-57. doi: 10.1007/s40135-013-0009-1. PMID 23710423
- [Background] Urzua CA, Vasquez DH, Huidobro A, Hernandez H, Alfaro J. Randomized double-blind clinical trial of autologous serum versus artificial tears in dry eye syndrome. Curr Eye Res. 2012 Aug;37(8):684-8. doi: 10.3109/02713683.2012.674609. Epub 2012 Jun 6. PMID 22670856
- [Background] Wolffsohn JS, Arita R, Chalmers R, Djalilian A, Dogru M, Dumbleton K, Gupta PK, Karpecki P, Lazreg S, Pult H, Sullivan BD, Tomlinson A, Tong L, Villani E, Yoon KC, Jones L, Craig JP. TFOS DEWS II Diagnostic Methodology report. Ocul Surf. 2017 Jul;15(3):539-574. doi: 10.1016/j.jtos.2017.05.001. Epub 2017 Jul 20. PMID 28736342
- [Result] Jeong, S. & Lee, S. B. 2016. Reliability of a New Non-Invasive Tear Film Break-up Time Measurement Using a Keratograph. Journal of the Korean Ophthalmological Society 57(9): 1354-1360.
- [Result] Mukhopadhyay S, Sen S, Datta H. Comparative role of 20% cord blood serum and 20% autologous serum in dry eye associated with Hansen's disease: a tear proteomic study. Br J Ophthalmol. 2015 Jan;99(1):108-12. doi: 10.1136/bjophthalmol-2013-304801. Epub 2014 Aug 19. PMID 25138758
- [Result] Rauz S, Koay SY, Foot B, Kaye SB, Figueiredo F, Burdon MA, Dancey E, Chandrasekar A, Lomas R. The Royal College of Ophthalmologists guidelines on serum eye drops for the treatment of severe ocular surface disease: full report. Eye (Lond). 2017 Nov 17. doi: 10.1038/eye.2017.209. Online ahead of print. No abstract available. PMID 29148532
- [Result] Rauz S, Saw VP. Serum eye drops, amniotic membrane and limbal epithelial stem cells--tools in the treatment of ocular surface disease. Cell Tissue Bank. 2010 Feb;11(1):13-27. doi: 10.1007/s10561-009-9128-1. Epub 2009 Apr 22. PMID 19387867
- [Result] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Result] Sharma N, Goel M, Velpandian T, Titiyal JS, Tandon R, Vajpayee RB. Evaluation of umbilical cord serum therapy in acute ocular chemical burns. Invest Ophthalmol Vis Sci. 2011 Feb 25;52(2):1087-92. doi: 10.1167/iovs.09-4170. PMID 20538982
- [Result] Simmons PA, Liu H, Carlisle-Wilcox C, Vehige JG. Efficacy and safety of two new formulations of artificial tears in subjects with dry eye disease: a 3-month, multicenter, active-controlled, randomized trial. Clin Ophthalmol. 2015 Apr 15;9:665-75. doi: 10.2147/OPTH.S78184. eCollection 2015. PMID 25931807
- [Result] Vajpayee RB, Mukerji N, Tandon R, Sharma N, Pandey RM, Biswas NR, Malhotra N, Melki SA. Evaluation of umbilical cord serum therapy for persistent corneal epithelial defects. Br J Ophthalmol. 2003 Nov;87(11):1312-6. doi: 10.1136/bjo.87.11.1312. PMID 14609821
- [Result] Versura P, Buzzi M, Giannaccare G, Terzi A, Fresina M, Velati C, Campos EC. Targeting growth factor supply in keratopathy treatment: comparison between maternal peripheral blood and cord blood as sources for the preparation of topical eye drops. Blood Transfus. 2016 Mar;14(2):145-51. doi: 10.2450/2015.0020-15. Epub 2015 Jul 9. PMID 26192781
- [Result] Yoon KC, Heo H, Im SK, You IC, Kim YH, Park YG. Comparison of autologous serum and umbilical cord serum eye drops for dry eye syndrome. Am J Ophthalmol. 2007 Jul;144(1):86-92. doi: 10.1016/j.ajo.2007.03.016. Epub 2007 May 9. PMID 17493572
- [Result] Yoon KC, Im SK, Park YG, Jung YD, Yang SY, Choi J. Application of umbilical cord serum eyedrops for the treatment of dry eye syndrome. Cornea. 2006 Apr;25(3):268-72. doi: 10.1097/01.ico.0000183484.85636.b6. PMID 16633024